CLINICAL TRIAL: NCT03032003
Title: Prophylactic Use of Cranberries in Recurrent Bacterial Cystitis in Women: A Randomized, Comparative, Study.
Brief Title: Prophylactic Use of Cranberries in Recurrent Bacterial Cystitis in Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Vasileios Tzortzis, Associated Professor, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cranberries1
Record Dates: First submitted 2017-01-13; First posted 2017-01-26 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Recurrent Urinary Tract Infections in Women
MeSH Terms: interventions — Cysticlean

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cysticlean arm (Active Comparator): Cysticlean (2 BID for 15 days)
  Interventions: Other: Cysticlean
- Placebo arm (Placebo Comparator): Placebo (2 BID for 15 days)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Cysticlean — 2 BID for 15 days
  Arms: Cysticlean arm
Other: Placebo — 2 BID for 15 days
  Arms: Placebo arm

SUMMARY:
To investigate if oral administration of 240mg PAC of cranberries can reduce the number of episodes of acute bacterial cystitis and improve general QoL in women with recurrent bacterial cystitis. In addition, the effect on vagina and rectal flora will studied and the adverse effect profile of the drug will be reported.

Women with ≥3 symptomatic episodes of lower UTIs at the previous year will be recruited from the outpatient population who present to their family physician or specialist with symptomatic recurrent UTI. Informed consent will be obtained from all patients and they will be divided in groups according to their age. Urinary culture, vaginal and rectal swab will be taken from all the patients. Antibiotic treatment will be prescribed (using the drug of choice according to the urine culture and the treating physician choice). Subsequently, they will be randomized to receive combined antibiotic treatment with one capsule of Cysticlean 240mg PAC two times per day or antibiotic treatment with placebo. At 14th day post treatment and after a negative urinary culture patients will continue to receive per os, daily, one capsule of Cysticlean 240mg at bed time for 12 months or placebo respectively.

Study visits will occur at 3rd, 6th , 9th and 12th month treatment phase. A urine collection, vaginal swabs and rectal swab will be taken at study entry and at the month 3, 6, 9 and 12 visits.

Participants will be asked about medication usage, any side effects they may be experiencing at each study visit. If participants develop a UTI at any time during the study, they will be asked to visit the study site within 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Negative urine culture
* At least 3 UTI's within 12 months prior to study entry

Exclusion Criteria:

* Anatomic abnormalities of the urinary tract
* Use of investigational drugs within 30 days prior to study entry
* Current use of warfarin
* Allergy or intolerance of cranberry products
* > 50 ml of residual urine (measured by US)
* Use of indwelling catheter
* uncontrolled diabetes
* creatinine > 250 mmol/l,
* Symptomatic vaginitis
* Pregnant or breastfeeding

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2017-02-15 (Estimated); Primary Completion 2018-03-31 (Estimated); Study Completion 2018-05-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of the use of Cranberries in the prevention of the recurrent UTIs is women. | 12 months
  Follow up with urinary cultures will be evaluated for Cranberries affection in UTIs

REFERENCES:
- [Derived] Tsiakoulias E, Gravas S, Hadjichristodoulou C, Oikonomou KG, Kyritsi M, Dadouli K, Matziri A, Kola K, Vacthsioli E, Tsiakoulia M, Gianniou M, Tzortzis V. Randomized, placebo-controlled, double-blinded study of prophylactic cranberries use in women with recurrent uncomplicated cystitis. World J Urol. 2024 Jan 12;42(1):27. doi: 10.1007/s00345-023-04741-0. PMID 38214795